CLINICAL TRIAL: NCT06531343
Title: Advancing Lung Cancer Screening: Artificial Intelligence, Multimodal Imaging and Cutting-Edge Technologies for Early Detection and Characterization
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Fondazione Policlinico Universitario Campus Bio-Medico (Other); University of Calabria (Other); University of Salerno (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Principal Investigator, IRCCS San Raffaele
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: PNRR-MCNT2-2023-12377755
Record Dates: First submitted 2024-07-23; First posted 2024-08-01 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-07

CONDITIONS: Lung Cancer Screening

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LDCT scan and simultaneous [18F]FDG PET/CT on new-generation long axial field of view scanner (Experimental)
  Interventions: Procedure: LDCT scan and simultaneous [18F]FDG PET/CT on new-generation long axial field of view scanner
- low LDCT only (Active Comparator)
  Interventions: Procedure: LDTC only

INTERVENTIONS:
Procedure: LDCT scan and simultaneous [18F]FDG PET/CT on new-generation long axial field of view scanner — 18F]FDG will be injected intravenously, and PET/CT images will be acquired after 60 minutes (± 10 minutes). PET/CT images will be first analysed with the lung window to detect any findings suggestive of a lung tumour.
  Whole-body PET/CT images will be then analysed to detect any incidental finding in the chest as well as other anatomical areas included in the field of view. PET/CT images will be considered positive if there is at least one non-calcified lung nodule or any suspicious finding on CT scan characterised by focal [18F]FDG uptake deviating from physiological distribution or above physiological background activity.
  Arms: LDCT scan and simultaneous [18F]FDG PET/CT on new-generation long axial field of view scanner
Procedure: LDTC only — The LDCT scan will be performed in single deep inspiratory breath hold. No intravenous contrast will be administered.
  Arms: low LDCT only

SUMMARY:
Currently available screening programmes for lung cancer are limited by many challenges including low diagnostic accuracy, radiation exposure and high costs. New technologies in PET/CT scanners can allow cheaper and more sensitive exams with low radiation exposure. AI can be used to denoise LDCT to enhance the accuracy of imaging tests and build riskassessment models. This project aims to develop a new approach exploiting both these revolutionary advancements to bridge the existing gap in lung cancer screening. Patients in a high-risk population will be enrolled into two different cohorts undergoing LDCT scan and simultaneous [18F]FDG PET/CT on new-generation long axial field of view scanner (UO1) or screening with low LDCT only (UO2). AI will assist in image enhancement and interpretation and will develop a personalised risk-model guiding the following steps of clinical management, significantly improving early diagnosis of lung cancer, reducing mortality and healthcare costs.

DETAILED DESCRIPTION:
Assessment of the potential added value of low dose [18F]FDG PET/CT in the early detection of lung cancer in the screening work-up of the high-risk population. The target population (cohort 1) for the multimodal screening programme will be identified at UO1 on the basis of the PLCOM2012 prediction risk model. All patients enrolled in cohort 1 will undergo a LDCT and a simultaneous low dose [18F]FDG PET scan. Whole body [18F]FDG PET/CT will be performed according to EANM Guidelines for tumour imaging. Briefly, patients will be instructed to fast for 6 hours and to avoid strenuous physical activity for 48 hours prior to the PET/CT scan. Diabetic patients will be instructed to fast for 4 hours prior to the scan and will be instructed on the use of medications according to the institution's protocol. Blood glucose levels will be checked, [18F]FDG will be injected intravenously, and PET/CT images will be acquired after 60 minutes (± 10 minutes). A new generation long axial field of view PET/CT scanner (Omni Legend, General Electric Healthcare, Waukesha, WI, USA) will be used for whole body imaging.

The control population (cohort 2) will be identified in UO2 on the basis of the PLCOM2012 prediction risk model as previously described for cohort 1. The LDCT scan will be performed in single deep inspiratory breath hold. No intravenous contrast will be administered. LDCT images will be assessed and interpreted by at least two experienced radiologists. LDCT will be defined as positive if at least one non-calcified lung nodule >5 mm in any diameter is detected. LDCT will be defined as negative if no clinically significant morphological alterations are detected. Non-calcified nodules of 3-5mm detected by LDCT will be reported. Lung-RADS criteria will be used to classify detected lung nodules. Any other suspicious morphological alteration will be reported. The number, size, characteristics, and location of any lesion detected will be recorded for each LDCT scan. Any abnormality suggestive of clinically significant conditions other than cancer will be also reported. Sensitivity, specificity, and accuracy will be calculated by per-patient and per-lesion analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years
* PLCOm2012 risk prediction > 4%
* Be willing to adhere to the study intervention through [18F]FDG PET/CT or LDCT imaging
* Signed written informed consent form

Exclusion Criteria:

* Blood glucose levels >200 mg/dl,
* Ongoing pregnancy and breastfeeding
* Unwillingness to participate,
* Previous diagnosis of lung cancer,
* Previous CT scan within the last 24 months
* Concomitant severe clinical conditions and any condition that preclude the feasibility of the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to assess the diagnostic accuracy of low-dose [18F]FDG PET/CT for screening in high-risk individuals or lung cancer Time Frame: | 24 months
  The primary endpoint is the detection rate of [18F]FDG PET/CT for suspicious lung nodules. The sensitivity, specificity and accuracy will be calculated by a per-patient and per-lesion analysis based on the clinico-radiological follow-up.
  PET/CT images will be considered positive if there is at least one non-calcified lung nodule or one suspicious finding on CT scan characterised by focal [18F]FDG uptake that deviates from the physiological distribution or is above the physiological background activity. If there are no areas of increased uptake compared to physiological background activity, PET/CT images are considered negative.

SECONDARY OUTCOMES:
Assessment of the diagnostic accuracy of LDCT alone for screening in high-risk individuals or lung cancer and accuracy of [18F]FDG PET/CT for the additional detection of non-lung cancers in a high-risk population. | 24 months
  The sensitivity, specificity and accuracy will be calculated by a per-patient and per-lesion analysis based on the clinico-radiological follow-up. LDCT will be defined as positive if at least one non-calcified lung nodule >5 mm in any diameter is detected. LDCT will be defined as negative if no clinically significant morphological alterations are detected. Lung-RADS criteria will be used to classify detected lung nodules.
  PET/CT images will be considered positive if there is at least one suspicious morphological finding on CT scan characterised by focal [18F]FDG uptake that deviates from the physiological distribution or is above the physiological background activity. If there are no areas of increased uptake compared to physiological background activity, PET/CT images are considered negative.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs San Raffaele, Milan, Italy